CLINICAL TRIAL: NCT04475055
Title: Reliability and Validity of the DIPS (Diagnostisches Interview Bei Psychischen Störungen; a Structured Interview to Assess Psychological Disorders) in a Community Sample
Brief Title: Reliability and Validity of the DIPS (Structured Interview) in a Community Sample
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Ruth von Brachel, Principal Investigator, Ruhr University of Bochum
Other Study IDs: 2014-149
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Psychological Disease
Keywords: clinical interview; community sample

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community sample: Participants will take part in the DIPS-interview and in an online survey.
  Interventions: Diagnostic Test: Diagnostisches Interview bei psychischen Störungen (DIPS)

INTERVENTIONS:
Diagnostic Test: Diagnostisches Interview bei psychischen Störungen (DIPS) — The DIPS is a structured interview which assesses the most frequent psychological disorders. It can be delivered by trained clinicians and takes between 50-120 minutes. Its acceptance with patients is very good.

SUMMARY:
The DIPS (Diagnostisches Interview bei psychischen Störungen) is a structured interview to assess a variety of the most frequent psychological disorders. Its reliability and validity has been studied in clinical samples. Since structured interviews are also used in non-clinical samples like epidemiological research the investigators would like to conduct a study in a community sample to test the interview's reliability, validity and acceptance.

DETAILED DESCRIPTION:
The DIPS (Diagnostisches Interview bei psychischen Störungen) is a structured interview to assess a variety of the most frequent psychological disorders. Its reliability and validity has been demonstrated in clinical samples. Also, studies have tested patients' and therapist's acceptance of the interview. Since structured interviews are also used in non-clinical samples like epidemiological research the investigators would like to conduct a study in a community sample to test the interview's reliability, validity and acceptance in this population (study aim 1). The investigators also plan to compare positive mental health and affective styles of the subsample of participants with no current or lifetime mental health illness to patients from the local outpatient treatment center at the Ruhr-University Bochum, who all reported at least one current mental illness (study aim 2). If the researchers obtain enough participants with no current mental health problem, but a history of at least one mental health illness, they will be included in the analysis for study aim 2 as well.

Since the data collection takes place during the Corona pandemic, participants will also be asked to give information about how they are affected, about their living situation and their media use over the course of half a year to describe the sample and to determine the impact of these factors on the incidence and course of mental illness (study aim 3).

ELIGIBILITY:
Inclusion Criteria:

* sufficient knowledge of the German language

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults who are willing to complete the structured interview and the questionnaires of the online-survey are allowed to take part in the study.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Affective Styles Questionnaire (ASQ, Hofmann & Kashdan, 2010) | Baseline
  A 20-item scale measuring the three affective styles concealing, adjusting, and tolerating, on a 5-point Likert scale ranging from (1) = "not true of me at all" to (5) = "extremely true of me". Higher scores indicate a stronger tendency towards concealing, adjusting and tolerating respectively.
Affective Styles Questionnaire (ASQ, Hofmann & Kashdan, 2010) | after 4 months
  A 20-item scale measuring the three affective styles concealing, adjusting, and tolerating, on a 5-point Likert scale ranging from (1) = "not true of me at all" to (5) = "extremely true of me". Higher scores indicate a stronger tendency towards concealing, adjusting and tolerating respectively.
Affective Styles Questionnaire (ASQ, Hofmann & Kashdan, 2010) | after 6 months
  A 20-item scale measuring the three affective styles concealing, adjusting, and tolerating, on a 5-point Likert scale ranging from (1) = "not true of me at all" to (5) = "extremely true of me".Higher scores indicate a stronger tendency towards concealing, adjusting and tolerating respectively.
Depression Anxiety Stress Scale -21 (DASS-21; Nilges et al., 2015) | baseline
  The DASS-21 is a 21-item scale that measures the negative emotional states of depression, anxiety, and stress on a 4- point severity/ frequency scale with higher scores indicating more severe depression, stress, and anxiety respectively.
Depression Anxiety Stress Scale -21 (DASS-21; Nilges et al., 2015) | after 1 month
  The DASS-21 is a 21-item scale that measures the negative emotional states of depression, anxiety, and stress on a 4- point severity/ frequency scale with higher scores indicating more severe depression, stress, and anxiety respectively.
Depression Anxiety Stress Scale -21 (DASS-21; Nilges et al., 2015) | after 2 months
  The DASS-21 is a 21-item scale that measures the negative emotional states of depression, anxiety, and stress on a 4- point severity/ frequency scale with higher scores indicating more severe depression, stress, and anxiety respectively.
Depression Anxiety Stress Scale -21 (DASS-21; Nilges et al., 2015) | after 3 months
  The DASS-21 is a 21-item scale that measures the negative emotional states of depression, anxiety, and stress on a 4- point severity/ frequency scale with higher scores indicating more severe depression, stress, and anxiety respectively.
Depression Anxiety Stress Scale -21 (DASS-21; Nilges et al., 2015) | after 4 months
  The DASS-21 is a 21-item scale that measures the negative emotional states of depression, anxiety, and stress on a 4- point severity/ frequency scale with higher scores indicating more severe depression, stress, and anxiety respectively.
Depression Anxiety Stress Scale -21 (DASS-21; Nilges et al., 2015) | after 5 months
  The DASS-21 is a 21-item scale that measures the negative emotional states of depression, anxiety, and stress on a 4- point severity/ frequency scale with higher scores indicating more severe depression, stress, and anxiety respectively.
Depression Anxiety Stress Scale -21 (DASS-21; Nilges et al., 2015) | after 6 months
  The DASS-21 is a 21-item scale that measures the negative emotional states of depression, anxiety, and stress on a 4- point severity/ frequency scale with higher scores indicating more severe depression, stress, and anxiety respectively.
Positive Mental Health Scale (PMH; Lukat et al., 2016) | baseline
  A brief 9-item scale that assesses positive mental health on a 4-point likert scale. Higher scores indicating positive mental heath.
Positive Mental Health Scale (PMH; Lukat et al., 2016) | after 4 months
  A brief 9-item scale that assesses positive mental health on a 4-point likert scale. Higher scores indicating positive mental heath.
Positive Mental Health Scale (PMH; Lukat et al., 2016) | after 6 months
  A brief 9-item scale that assesses positive mental health on a 4-point likert scale. Higher scores indicating positive mental heath.
Acceptance of the interview (Bruchmüller et al., 2009) | after 4 months (after the interview)
  A 10-item scale that assesses the participants acceptance of the DIPS on a 5-point likert scale. Higher scores indicate higher acceptance.

SECONDARY OUTCOMES:
Family Climate Scale (FCS) | Baseline
  The FCS is a multilevel, self-report, whole-family index of aspects of family culture and process for use in nonclinical settings with families where the children may be adults. The questionnaire consists of a 60- items (10- items per subscale) on a ﬁve-point Likert-type responseformat, each including at least four reverse-codeditems, to guard against response set. Higher Scores indicate better family functioning.
Therapeutisch Relevante Belastungsliste (TRB; reasons for therapy) | after 4 months (after the interview)
  A 29- Item scale assessing the reasons behind a participants wish to receive psychotherapy. Higher scores indicate a higher need for therapy.
The Fear Questionnaire - Der Angstfragebogen (FQ; Hank et al., 1990) | after 4 months (after the interview)
  A 15- item questionnaire measuring the extent to which specific situations are avoided in order to measure the level of anxiety. Higher scores indicate more severe avoidance/ fear .
The Agoraphobia Cognitions Questionnaire (ACQ; Ehlers et al., 1993), | after 4 months (after the interview)
  A 15- item questionnaire that assesses fear related cognitions. Higher scores indicate higher levels of fear related cognitions.
Mobility Inventory for Agoraphobia (MI; Chambless et al., 1985) | after 4 months (after the interview)
  A 27-item inventory for the measurement of self-reported agoraphobic avoidance behavior and frequency of panic attacks with higher scores indicating more severe avoidance and a higher frequency of panic attacks.
Body Sensations Questionnaire (BSQ; Chambless et al., 1984), | after 4 months (after the interview)
  A 17-item questionnaire to measure the extent of anxiety in psychosomatic or functional complaints and non-organic somatic symptoms. A 5-point scale is used to assess the extent to which the symptom in question is causing fear or worry with 5 indicating more severe worries/ sensations.
Beck-Depression-Inventory-II (BDI-II; Hautzinger et al., 2006) | after 4 months (after the interview)
  A 21-question multiple-choice self-report inventory for measuring the severity of depression. Each answer is being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms
Fragebogen zu Gedanken und Gefühlen (FGG; questionnaire assessing thoughts and feelings; Renneberg et al., 2010) | after 4 months (after the interview)
  A 14- item screening tool for borderline-specific thinking. A high value is synonymous with a high level of approval for the individual items of the FGG.
Suicidal Behaviors Questionnaire-Revised (SBQ; Osman et al., 2001) | after 4 months (after the interview)
  The SBQ-R is designed to identify risk factors for suicide. Its based on four questions. A total score of 7 and higher in the general population and a total score of 8 and higher in patients with psychiatric disorders indicates significant risk of suicidal behavior.
Eating Disorder Examination Questionnaire (EDE-Q; Mond et al., 2006) | after 4 months (after the interview)
  The 28- item questionnaire is designed to assess eating disorder psychopathology. The EDE-Q is scored using a 7-point, forced-choice rating scale (0-6) with scores of 4 or higher indicative of clinical range.
Exzessives Computerspielen und Computerspielabhängigkeit im Jugendalter (excessive video game playing and video game addiction in adolescence; KFN-CSAS-II; Rehbein et al., 2009)) | after 4 months (after the interview)
  A14- item questionnaire, that assesses online gaming behaviour. A total value is determined for all items with which the severity of the symptom burden can be assessed.
LAST - Lübecker Alkoholabhängigkeit- und -missbrauch-Screening-Test (screening for alcohol dependency and abuse; Rumpf et al., 2001) | after 4 months (after the interview)
  The last is a short, sensitive screening test for the detection of alcohol addiction and abuse. It contains 7 items, to be answered with "yes" or "no". A sum of 2 or more points indicates alcohol abuse or alcohol addiction.
Penn State Worry Questionnaire (PWQ; Glöckner-Rist et al., 2014) Penn State Worry Questionnaire (PSWQ) | after 4 months (after the interview)
  A 16-item questionnaire, that identifies excessive, unrealistic worries as the central cognitive syndrome of generalized anxiety disorder.Items are rated on a five-point scale: 1-Not at all typical of me to 5-Very typical of me. Possible range of scores is 16-80 with the algorithm of total scores: 16-39 low worry, 40-59 moderate worry, and 60-80 high worry.
State-Trait Anxiety Inventory (STAI; Spielberger et al., 1994). | after 4 months (after the interview)
  Its an inventory based on a 4-point Likert scale and consists of 40 questions measuring state and trait anxiety. Higher scores indicate greater anxiety.
Whiteley-Index (WI; Hinz et al., 2003) | after 4 months (after the interview)
  An instrument for measuring hypochondria. Hypochondrical worries and beliefs are assessed with 14 items with higher scores indicating more severe hypochondria.
Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 1989) | after 4 months (after the interview)
  The PSQI measures sleep quality on a 10-item scale.Higher scores indicate worse sleep quality.
PTSD Checklist for DSM-5 (PCL-5; Belvins et al., 2015) | after 4 months (after the interview)
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. A provisional PTSD diagnosis can be made by treating each item rated as 2 = "Moderately" or higher as a symptom endorsed, then following the DSM-5 diagnostic rule which requires at least: 1 B item (questions 1-5), 1 C item (questions 6-7), 2 D items (questions 8-14), 2 E items (questions 15-20).
Symptom Checklist-90-R (SCL-90-R; Hessel et al., 2001) | after 4 months (after the interview)
  Nine scales (10 questions per scale) (somatization, compulsiveness, insecurity in social contact, depression, anxiety, aggressiveness / hostility, phobic anxiety, paranoid thinking, psychoticism) and three global parameters (GSI, PSDI, PST) assess the psychological stress in the past seven days. It is scored on a five-point Likert scale, indicating the rate of occurrence of the symptom during the time reference. Higher scores indicate more severe symptoms.
Balanced Inventory of desireable Responding (BIDR; Paulhus; 1991) | after 4 months (after the interview)
  The questionnaire consists of two scales with 10 items each measuring two aspects of social desirability: self- deceptive enhancement and impression management. On a 7-point likert scale (from "1 = does not apply at all" to "7 = applies fully") it is assessed to what extent participants agree or disagree with the statements with higher scores representing social desirability.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Schneider, Prof., Study Director — Ruhr-University Bochum
Locations (1):
- Ruhr-University, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided